CLINICAL TRIAL: NCT01110824
Title: Prevention of Left Ventricular Dysfunction With Enalapril and Carvedilol in Patients Submitted to Intensive Chemotherapy for the Treatment of Malignant Hemopathies
Brief Title: Prevention of Left Ventricular Dysfunction During Chemotherapy
Acronym: OVERCOME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); European Union (Other)
Responsible Party: Principal Investigator, Xavier Bosch, Dr., Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OVERCOME; 2007-006604-38 (EudraCT Number); FIS EC07/90211 (Other Grant/Funding Number: ISCIII)
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Acute Myeloid Leukemia; Precursor-cell Lymphoblastic Leukemia-Lymphoma; Lymphoid Neoplasm; Multiple Myeloma; Lymphoma; Autologous Hematopoietic Stem Cell Transplantation
Keywords: Prevention; ventricular dysfunction; chemotherapy; acute myeloid leukemia; precursor-cell lymphoblastic leukemia; multiple myeloma; lymphoma; ejection fraction; Autologous hematopoietic stem cell transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Multiple Myeloma; Lymphoma; Ventricular Dysfunction | interventions — Enalapril; Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enalapril and carvedilol (Experimental): Enalapril 2.5 to 10 mg BID plus Carvedilol 6.25 to 25 mg BID
  Interventions: Drug: Enalapril and carvedilol
- Control (No Intervention): Control arm without intervention

INTERVENTIONS:
Drug: Enalapril and carvedilol — Enalapril 2.5 to 10 mg BID Carvedilol 6.25 to 25 mg BID
  Arms: Enalapril and carvedilol

SUMMARY:
The investigators' objective is to assess the efficacy of the combined treatment with enalapril and carvedilol in the prevention of left ventricular systolic dysfunction in patients with hematological malignancies submitted to intensive chemotherapy with potential cardiotoxicity.

The hypothesis is that these drugs administered during chemotherapy may prevent left ventricular systolic dysfunction.

DETAILED DESCRIPTION:
The prognosis of patients with hematological malignancies has greatly improved in the last years with the use of new chemotherapeutic drugs and regimens at the cost of significant adverse events such as cardiac toxicity. Asymptomatic left ventricular systolic dysfunction limits the specific treatment of the patients and their long-term survival, since a significant proportion of them will relapse within 5 years after front-line therapy and will require further salvage treatment, including hematopoietic stem-cell transplantation in most instances.

Angiotensin-converting enzyme inhibitors (ACEIs) have showed to have preventive effects against chemotherapy-induced cardiotoxicity in animal models, and in patients with early cardiotoxicity. Carvedilol prevent free radical release, mitochondrial dysfunction, apoptosis, and dilated cardiomyopathy in animals treated with anthracyclines, and have shown promising results in preventing chemotherapy-induced left ventricular dysfunction in patients.

As demonstrated in post-infarction patients, the combined treatment with an ACEI and carvedilol could have additive effects to prevent LV dysfunction in patients with hematological malignancies at high risk of cardiac toxicity. Therefore, we designed the OVERCOME (preventiOn of left Ventricular dysfunction with Enalapril and caRvedilol in patients submitted to intensive ChemOtherapy for the treatment of Malignant hEmopathies) study, a prospective, randomized trial to evaluate the combined effect of enalapril and carvedilol on the prevention of left ventricular dysfunction in patients with malignant hemopathies undergoing intensive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-70 years old
* Sinus rhythm
* Normal LVEF (>=50%)
* Patients recently diagnosed of acute leukemia to be submitted to intensive chemotherapy or
* Patients with other hemopathies submitted to autologous peripheral blood stem cell transplantation
* Signed informed consent

Exclusion Criteria:

* Congestive heart failure
* LVEF<50%
* Coronary artery disease,
* significant valvulopathy or myocardiopathy
* Renal failure (MDRD<30)
* Liver failure
* Ongoing or expected need to be treated with angiotensin-converting enzyme inhibitors (ACE-i),angiotensin II receptor blockers (ARB) or beta-blockers
* Prior allergy to ACEI or ARB
* Systolic blood pressure <90 mmHg
* Asthma
* Auriculoventricular (AV) block or sinus bradycardia (HR<60 bpm)
* Persistent atrial fibrillation
* Need to be treated with Class I antiarrhythmic drugs
* Pregnancy
* Inability or unwillingness to give unformed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-04; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in left ventricular ejection fraction (LVEF) measured by echocardiography and by cardiac magnetic resonance imaging (CMR). | 6 months after randomization

SECONDARY OUTCOMES:
Incidence of death, heart failure or LV systolic disfunction (LVEF<45%) | 6 months after randomization
Assessment of genetic polymorphisms involved in chemotherapy-induced cardiotoxicity | Baseline
Prognostic value for cardiac toxicity of troponin I and BNP | up to 3 months
Right and left ventricular volumes measured by CMR | 6 months after randomization
Subgroup analysis by diagnosis (acute leukemia vs. other malignant hemopathies submitted to autologous peripheral blood stem cell transplantation), and positive biomarkers (TnI, BNP). | 6 months after randomization
Incidence of an absolute decrease in LVEF>10 percent units associated with a decline below its normal limit of 50% | 6 months after randomization
Serious adverse events | 6 months after randomization
the incidence of LV dysfunction as assessed by the measurement of the LV strain, and of diastolic dysfunction measured by echo-Doppler | 6 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Bosch, M.D., PhD., Study Chair — Hospital Clinic, University of Barcelona
Locations (1):
- Hospital Clinic, Barcelona, Catalonia, Spain

REFERENCES:
- [Background] Bosch X, Esteve J, Sitges M, de Caralt TM, Domenech A, Ortiz JT, Monzo M, Morales-Ruiz M, Perea RJ, Rovira M. Prevention of chemotherapy-induced left ventricular dysfunction with enalapril and carvedilol: rationale and design of the OVERCOME trial. J Card Fail. 2011 Aug;17(8):643-8. doi: 10.1016/j.cardfail.2011.03.008. Epub 2011 May 6. PMID 21807325
- [Result] Bosch X, Rovira M, Sitges M, Domenech A, Ortiz-Perez JT, de Caralt TM, Morales-Ruiz M, Perea RJ, Monzo M, Esteve J. Enalapril and carvedilol for preventing chemotherapy-induced left ventricular systolic dysfunction in patients with malignant hemopathies: the OVERCOME trial (preventiOn of left Ventricular dysfunction with Enalapril and caRvedilol in patients submitted to intensive ChemOtherapy for the treatment of Malignant hEmopathies). J Am Coll Cardiol. 2013 Jun 11;61(23):2355-62. doi: 10.1016/j.jacc.2013.02.072. Epub 2013 Apr 10. PMID 23583763